CLINICAL TRIAL: NCT00308074
Title: A Prospective Open-Label Trial of Aripiprazole Monotherapy in the Autism Spectrum Disorders (ASD)
Brief Title: An Open-Label Trial of Aripiprazole in Autism Spectrum Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Jean Frazier, Director, Child & Adolescent Neuropsychiatric Research Program, Cambridge Health Alliance
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-0119/06/05
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Autism; Asperger's Disorder; Pervasive Developmental Disorder
Keywords: behavioral problems; aggression; autism; aripiprazole
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive; Problem Behavior; Aggression | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole (Experimental): aripiprazole monotherapy, begun at 2.5 mg or 5.0 mg based on clinical impression and severity of aggression and agitation. Dose to be adjusted in not more than 5 mg increments, weekly. The lowest effective dose will be used up to a maximum daily dose of 20 mg.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — open-label, flexible-dosing
  Other Names: Abilify

SUMMARY:
The aim of this study is to evaluate the efficacy, safety and tolerability of aripiprazole monotherapy in the treatment of children and adolescents suffering from Autism Spectrum Disorder (ASD) over a 12-week period. We hypothesize that aripiprazole may be helpful in reducing ASD-associated symptoms of anxiety and aggression, resulting in significant improvements in global outcome.

DETAILED DESCRIPTION:
Study Design: Fifteen patients with DSM-IV diagnoses of Autism, Asperger's Disorder or Pervasive Developmental Disorder Not Otherwise Specified (PDD NOS) will be enrolled in this 12-week open-label study. Parents of potential subjects will do a preliminary phone screen, followed by a clinical evaluation by a psychiatrist for possible inclusion in the study. Informed written consent and assent will be obtained from the parents and subjects respectively once deemed competent and before the initiation of any study procedures.

Clinical Evaluation will use the Autism Diagnostic Interview (ADI-R) and the Autism Diagnostic Observation Schedule (ADOS) to establish a formal diagnosis.

Study Procedures Baseline Assessments: Many baseline measures for physical health will be done at the screening visit and during the first weekly visit. These will include a clinical interview, physical and neurological examination will be done during the screening period and height, weight and vital signs, and a calculation of his/her Body Mass Index (BMI) will be done during the screening period and during the first weekly visit. Laboratory measures at baseline and study completion will include a complete metabolic panel (with liver transaminases) and complete blood count with differential. Further measures will include a fasting lipid profile, hemoglobin A1C, prolactin level and insulin levels, and fasting blood sugar level (FBS). Serum albumin will be measured not only as a measure of nutritional state, but also in accordance with the fact that aripiprazole is 99% protein-bound. An electrocardiogram (ECG) will be performed at the beginning and end of the study to monitor for possible cardiac effects. These measures are aimed at monitoring side effects reported in the use of other medications in this class. Urine pregnancy tests will be performed for each female subject at the beginning and end of the study.

Outcome measures will include the Yale-Brown Obsessive Compulsive Scale (Y-BOCS), Brief Psychiatric Rating Scale for children (BPRS-C), Clinical Global Impression - Severity (CGI-S), Vineland Adaptive Behavior Scale (VABS) and the Atypical Children's Development Scale (ACDS).

Baseline parameters for extrapyramidal side effects will be established using the Abnormal Involuntary Movement Scale (AIMS), the Simpson Angus Extrapyramidal Side Effect Scale (SAEPS) and the Barnes Akathisia Rating Scale. Baseline values for general side effects will be compiled using the Monitoring of Side Effects System (MOSES).

Weekly visits: At all visits, patients will undergo a clinical interview, vital signs, and weight measures. Custodial guardian(s) will provide collateral information. The weekly "short" visits will occur at weeks 2, 4, 6, 8, 10 and 12. They will be about 45 minutes in duration.

Ongoing outcome measures will be performed at visits 3, 5, 7, 9 and 11. The visits will be about 1-1.5 hours in duration. The measures done will include those at the short visits, as well as the Y-BOCS, BPRS, ABC and CGI-S. Side effects will be monitored using the AIMS, SAEPS, Barnes Akathisia Scale and MOSES at these visits.

Termination Visit: The last visit (Visit 13 or earlier if patient drops out of the study) will include the repetition of all measures at visit 1 (except the ADI-R) and will last about 2 hours. All baseline laboratory measures will be repeated at this time.

Follow-Up Patient Care: After completion of the clinical trial, the patients will be followed at the Cambridge Health Alliance (CHA) Center for Child and Adolescent Development until they can be referred back to their original psychiatric providers or to appropriate treatment providers in the community.

Medication dosing: Aripiprazole will be started at 2.5mg or 5mg depending on clinical impression and severity of especially aggression and agitation. At the weekly visits, the dose will be adjusted in not more than 5mg increments according to clinical impression. The lowest effective dose will be used, up to a maximum dose of 20mg.

Patients already taking psychotropic medications will be tapered off their medications during the first 1-2 weeks of the study. The dose will be reduced to 67% of the initial dose for 3 days and then to 33% of the initial dose for 3 days and then the medication(s) will be discontinued. The subjects will remain off of on enrollment medications for 5 half lives and then aripiprazole will be initiated. Anticonvulsant medications taken for seizure control may be continued throughout the trial as long as the subject has been on a stable dose for 30 days prior to the study and has been seizure free for 6 months. These medication doses will be held stable throughout the trial.

Adverse Events: Any serious adverse event leading to hospitalization will lead to study discontinuation. Any event requiring concomitant medication(s) will also lead to discontinuation. Adverse events will be reported to the Institutional Review Board (IRB) if there is an event requiring medical attention, or scores 3 or higher on the MOSES scale. Also, failure to comply with the study instructions will result in termination from the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females ages 6-17
* A diagnosis of Autism, Asperger's Disorder, or Pervasive Developmental Disorder - not otherwise specified (PDD NOS)
* Medically healthy
* Ability to give assent
* Significant tantrums, aggression, self-injurious behavior and/or agitation by achieving a score of 18 or higher on the Aberrant Behavior Checklist-irritability subscale and a score of moderate or higher on the Clinical Global Impressions-Severity Scale.

Exclusion Criteria:

* Co-morbid serious mental illness.
* Intelligence Quotient (IQ) <50, based on verified records of cognitive testing performed within 2 years of enrollment. In event that suitable records of prior testing are unavailable, IQ will be estimated using the Wechsler Abbreviated Scale of Intelligence (WASI, 1999 Harcourt Assessment, Inc.).
* Significant active medical and/or neurological illness.
* Subjects that require other psychotropic medications such as antidepressants, mood stabilizers, anticonvulsants, stimulants, sedatives, or other antipsychotic medications in order to maintain clinical stability.
* Active substance abuse/dependence based upon history and urine toxicology screen.
* Inability to have blood drawn at baseline and termination visits.
* Known allergy or hypersensitivity to aripiprazole or its ingredients.
* Patients clinically stable on current medications.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean A Frazier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Medford, Massachusetts, United States

REFERENCES:
- See also: Research program website — http://www.challiance.org/research/research.shtml

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment will take place from mainly the Cambridge Health Alliance clinics, and the McLean Hospital affiliated service site for children and adolescents with an autism spectrum disorder (ASD), but also from other healthcare facilities in the vicinity.
Pre-assignment Details: All individuals enrolled will have Diagnostic and Statistical Manual Fourth Edition (DSM-IV) diagnoses of Autism, Asperger's Disorder or Pervasive Developmental Disorder, not otherwise specified (PDD NOS) and will be enrolled in this 12-week open-label study
Groups:
- Aripiprazole: aripiprazole monotherapy
  Aripiprazole will be started at 2.5 or 5mg depending on clinical impression and severity of aggression and agitation. The dose will be evaluated weekly, according to clinical impression and adjusted if deemed appropriate, in not more than 5mg increments . The lowest effective dose will be used.
Period: Overall Study
Arm/Group | Aripiprazole
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Aripiprazole: aripiprazole monotherapy
Arm/Group | Aripiprazole
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13 (1.66)
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impressions-Improvement
Description: The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to evaluate how much the patient's illness has improved or worsened compared to their baseline condition at the beginning of the intervention. The ratings are evaluated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: Baseline, Endpoint using last observation carried forward (LOCF) at weeks 3,5,7,9,11 and 13.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 14
units on a scale | 1.8 (1.6)

2. Primary Outcome: Aberrant Behavior Checklist-Irritability Subscale
Description: Aberrant Behavior Checklist (ABC) The ABC is a 58 item symptom checklist for assessing problem behaviors in individuals ages 6 to 54 with mental retardation. Items are rated on a 4-point scale (0=no problem to 3=severe problem). A decrease in score indicates improvement.
  There are five subscales: a) Irritability and Agitation b) Lethargy and Social Withdrawal c) Stereotypic Behavior d) Hyperactivity and Noncompliance and e) Inappropriate Speech.This study uses the Irritability subscale for its outcome. The Irritability subscale is the sum of 15 items. Each item is rated using the scale: 0 = Not at all; 1 = Slight in degree; 2 = Moderately serious; and 3 = Severe in degree. The Irritability subscale total score ranges from 0 to 45. A decrease in score over time indicates improvement.
Time Frame: Baseline, Endpoint using last observation carried forward (LOCF) at weeks 3,5,7,9,11 and 13.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 14
units on a scale
  Baseline irritability score | 24.5 (10.5)
  Endpoint irritability score | 8 (7.9)

3. Secondary Outcome: Yale-Brown Obsessive Compulsive Scale (Y-BOCS)
Description: 10-item assessment of obsessive-compulsive symptoms in patients less than 18 years of age. There are 5 items pertaining to compulsions rate symptoms (time spent, interference with functioning, distress, resistance, control) on a 5-point scale ( from 0=no symptoms/minimum severity, to 4=extreme symptoms/maximum severity). Total is the sum of 10 items. The range of possible totals is 0 (no symptoms) to 40 (severe). A decrease in value indicates improvement.
Time Frame: Baseline, Endpoint using last observation carried forward (LOCF) at weeks 3,5,7,9,11 and 13.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 14
units on a scale
  Baseline score | 15.9 (9.5)
  Endpoint score | 9.9 (6.9)

4. Secondary Outcome: Brief Psychiatric Rating Scale for Children (BPRS-C)
Description: The Brief Psychiatric Rating Scale for Children is a 21-item rating scale to evaluate psychiatric problems based on the clinician' s interview with the child/adolescent and parents. It has 7 scales: behavioral problems, depression, thought disorders, psychomotor excitation, withdrawal-retardation, anxiety, organicity. Ratings are based on a 7 point scale, from "Not Present" (scores 0) to "Extremely Severe" (scores 6 points). Total is the sum of the 21 items. The range of possible totals is 0 (no symptoms) to 126 (extremely severe).A decrease in score indicates improvement.
Time Frame: Baseline, Endpoint using last observation carried forward (LOCF) at weeks 3,5,7,9,11 and 13.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 14
units on a scale
  Baseline score | 69.0 (17.4)
  Endpoint score | 36.1 (14.9)

ADVERSE EVENTS:
Time Frame: 2 years, 10 months
Description: Labs, vital signs, ECG and the MOSES were collected at scheduled intervals.
Arm/Group | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=14)
neutropenia (Blood and lymphatic system disorders) | 1 (1) — Baseline -10 yo male no physical complaints; nausea,vomiting reported later in day. Baseline labs included WBC of 3500µl;absolute neutrophil 560. Study drug delayed for add'tl evaluation. Repeat CBC week later,results normal and throughout the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No